CLINICAL TRIAL: NCT02737540
Title: Neuropsychological Factors Associated With Vulnerability to Suicidal Behavior in Depressed Elderly Patients
Acronym: SPAD
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/MW-01
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major depressive episode: This study population consists of patients over 60 years of age with or without a personal history of suicide attempts, hospitalized in the Nîmes University Hospital psychiatry department or the Sophoras clinic for a major depressive episode.
- Healthy subjects: Healthy subjects over 60 years, not depressed and without personal history of severe mental illness or suicide attempts will be recruited.

SUMMARY:
The main objective of this study is to confirm the existence of risky decision making in a non strategic situation (Iowa Gambling Task) and a deficit of decision making in social situations, linked to greater sensitivity to injustice (Ultimatum Game) and a lower level of trust (Trust Game) in elderly depressed patients with a history of suicide attempts in comparison with older depressed patients without a history of suicidal acts and healthy subjects.

DETAILED DESCRIPTION:
The secondary objectives are to confirm or explore the deficits of certain cognitive processes involved in potentially suicidal behavior in depressed elderly persons but that have been little or not studied to date. These include:

A. cognitive control and sensitivity to interference (Victoria Stroop test, incompatibility test, flexibility test, Go / No-Go);

B. Strategic recovery of semantic memory (verbal fluency test);

C. Working memory (TEA);

D. Insight related to depression (Mood Disorders Insight Scale);

E. Recognition of facial emotions;

F. Emotional regulation;

G. Negative attitudes;

H. Self-perception and;

I. Time perspectives.

Finally, patients will be contacted by telephone at month 6 to assess the occurrence of a suicidal act during this period and thus calculate the predictive ability of cognitive and psychological factors.

ELIGIBILITY:
Inclusion criteria for patients:

* The patient or his/her representative must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patients with a diagnosis of current, moderate to severe, major depressive episode according to the DSM diagnostic criteria 5. This episode can be considered as part of a major depressive disorder or bipolar disorder.
* Patients with or without a personal history of suicide attempts. A suicide attempt is defined as any act performed with some intent to die (Mann 1998). Suicidal threats, aborted or interrupted gestures as well as self-mutilating acts without suicidal intent will not be considered as suicidal acts.
* Patients hospitalized (or followed as outpatients) in the Nîmes University Hospital psychiatry department or the Sophoras clinic in Nimes

Inclusion criteria for healthy subjects:

* The subject or his/her representative must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan
* Non-depressed subject without personal history of lifetime mood disorder or severe mental illness, or substance or alcohol abuse during the past 12 months

Exclusion criteria for patients:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient (or his/her legal representative) refuses to sign the consent
* It is impossible to correctly inform the patient or his/her legal representative
* The patient has a known MMSE score <24 (elimination of probable dementia pathology)
* Known central neurological disease including degenerative disease, severe head trauma and severe cerebral vascular disease
* Known schizophrenia and other psychotic disorders
* Alcohol or substance abuse in the last 12 months
* Electroconvulsive therapy in the 12 months preceding the study because of the risk of mnesic side effects
* Inability to perform neuropsychological tests because of a language problem, poor understanding, a major tremor, inability to sit still, a major sight problem that can not be corrected, or other severe cognitive impairment
* The subject presents an acute somatic decompensation incompatible with the completion of this study
* The patient has current confusion

Exclusion criteria for healthy subjects:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection
* The subject (or his/her legal representative) refuses to sign the consent
* It is impossible to correctly inform the subject or his/her legal representative
* The subject has a known MMSE score <24 (elimination of probable dementia pathology)
* Known central neurological disease including degenerative disease, severe head trauma and severe cerebral vascular disease
* Known schizophrenia and other psychotic disorders
* Alcohol or substance abuse in the last 12 months
* Electroconvulsive therapy in the 12 months preceding the study because of the risk of mnesic side effects
* Inability to perform neuropsychological tests because of a language problem, poor understanding, a major tremor, inability to sit still, a major sight problem that can not be corrected, or other severe cognitive impairment
* The subject has a mood disorder
* The subject presents an acute somatic decompensation incompatible with the completion of this study
* Thesubject has current confusion

Pharmacological treatment is not a criterion for exclusion in itself but it will be left to the judgment of the evaluator to choose to include a subject or not (or to postpone inclusion) depending on the drug (eg. after weaning daytime sedative treatment and benzodiazepines).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients over 60 years of age with or without a personal history of suicide attempts, hospitalized in the Nîmes University Hospital psychiatry department or the Sophoras clinic for a major depressive episode. Healthy subjects over 60 years, not depressed and without personal history of severe mental illness or suicide attempts will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Trust Game | Days 1-7
Ultimatum Game | Days 1-7
Iowa Gambling Task | Days 1-7

SECONDARY OUTCOMES:
Stroop Victoria Test | Days 1-7
Incompatibility Test | Days 1-7
Flexibility test | Days 1-7
Go-NoGo | Days 1-7
Working memory - TEA | Days 1-7
Mood Disorders Insight Scale | Days 1-7
Verbal fluency test | Days 1-7
Future autobiographical fluency task | Days 1-7
Bristol Emotion Recognition Test | Days 1-7
Cognitive Emotion Regulation Questionnaire | Days 1-7
Questionnaire on negative attitudes towards problems | Days 1-7
Revised self-awareness scale, Self-reference task | Days 1-7
Balanced Temporal Perspective Scale | Days 1-7
Suicide attempt within 6 months of follow-up | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice JOLLANT, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Clinique Les Sophoras, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Background] Mann JJ. The neurobiology of suicide. Nat Med. 1998 Jan;4(1):25-30. doi: 10.1038/nm0198-025. No abstract available. PMID 9427602